CLINICAL TRIAL: NCT03083015
Title: A Comparative Study Between Pulp Revascularization and MTA Apexification in Necrotic Immature Anterior Teeth, A Randomized Controlled Trial
Brief Title: Pulp Revascularization Versus MTA Apexification
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enas Ebrahim Sayed (Other)
Responsible Party: Sponsor-Investigator, Enas Ebrahim Sayed, Dentist at ministry of health, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Revas1; cebd (Other: center of evidence based/cu)
Record Dates: First submitted 2017-03-07; First posted 2017-03-17 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Necrotic Pulp
Keywords: regeneration, MTA apexification and TAP; revascularization
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Regeneration; Apexification

STUDY DESIGN:
Intervention Model Description: participants are allocated at random to receive one of two interventions according to the research plan. In RCT the outcomes are measured, so it is considered a quantitative study . This trial conforms to the Consolidated Standard of Reporting Trials (CONSORT)statement.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For the allocation concealment mechanism, each of 66 papers (each paper was eight folded) numbered from 1 to 66 were, individually packed, in opaque envelopes. Each participant picked an envelope at the beginning of the second visit. The number in the envelope determined which procedure was to be performed for the patient. The partner was to decide the procedure for the operator according to that number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revascularization (Experimental): Blood clot initiation and grey MTA ( Mineral Tri-oxide Aggregate) cervically compacted.
  Interventions: Procedure: revascularization
- Apexfication (Active Comparator): Apexification using grey MTA apically compacted without mechanical preparation.
  Interventions: Procedure: Apexification

INTERVENTIONS:
Procedure: revascularization — a sterile sharp needle was used to irritate the apical tissue until bleeding occurred apically in the root canal space so as to create a biological scaffold for the regenerative process
  Other Names: regeneration
  Arms: Revascularization
Procedure: Apexification — a 3-5 mm thickness of MTA using a hand plugger and was verified radiographically.
  Arms: Apexfication

SUMMARY:
This study compared the efficiency of pulp revascularization and MTA apexification in the treatment of patients with necrotic immature anterior teeth.

DETAILED DESCRIPTION:
the participants with 66 anterior necrotic immature teeth were randomly assigned into two equal groups with 33 teeth per each, according to regeneration and MTA apexification. At the first visit, all teeth were accessed and irrigated with NaOCl then a TAP was applied as intra-appointment intracanal medication. At the second visit, after removal of the medication with the irrigation, bleeding was initiated into the canal and isolated by the MTA in the orifice in the regeneration group. While in the Apexification group, the MTA was packed apically and all teeth were finally restored with resin composite restorations. The patients were recalled after 1, 3, 6, and 9 months for clinical and radiographic follow up.

ELIGIBILITY:
Inclusion Criteria:

* Medically-free patients having immature necrotic anterior teeth (with or without apical periodontitis/abscess) even with previous intervention.

Exclusion Criteria:

* History of allergy to any of the antibiotics in the tri-mix used in the study
* Patients with systemic diseases e.g. Diabetes mellitus, bleeding disorders,…
* Psychological disturbance
* External / internal root resorption or cystic lesion.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2015-12-02 (Actual); Study Completion 2015-12-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity measures | 2 days
  self reported pain intesity at 4, 12, 24, and 48 hours.(0= no pain and 100=worst pain) with a scale from 0 to 100 after the two visits.

SECONDARY OUTCOMES:
Resolution of periapical pathosis | 9 months
  Radiographically: by comparing radiolucencies in 9 months postoperative radiograph to the baseline radiograph.
Amount of radiographic increase in root length: | baseline and 9 months
  Root length was measured as a straight line from the cement-enamel junction to the radiographic apex of the tooth in millimeters = (9months follow up length - baseline length)
Amount of radiographic increase in the root dentinal wall thickness: | baseline and 9 months
  Dentin thickness was measured by =root thickness-pulp space and compared to the baseline radiograph measurements.
Decrease of apical diameter: | baseline and 9 months
  the diameter of the apical foramen was measured in millimeters and compared to the baseline radiograph measurements

CONTACTS AND LOCATIONS:
Overall Officials: ahmed alkhadem, lecturer, Principal Investigator — evidence based center, Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saoud TM, Zaazou A, Nabil A, Moussa S, Lin LM, Gibbs JL. Clinical and radiographic outcomes of traumatized immature permanent necrotic teeth after revascularization/revitalization therapy. J Endod. 2014 Dec;40(12):1946-52. doi: 10.1016/j.joen.2014.08.023. Epub 2014 Oct 16. PMID 25443280
- [Result] Alobaid AS, Cortes LM, Lo J, Nguyen TT, Albert J, Abu-Melha AS, Lin LM, Gibbs JL. Radiographic and clinical outcomes of the treatment of immature permanent teeth by revascularization or apexification: a pilot retrospective cohort study. J Endod. 2014 Aug;40(8):1063-70. doi: 10.1016/j.joen.2014.02.016. Epub 2014 Jun 13. PMID 25069909
- See also: test link — http://dx.doi.org/10.1016/j.joen.2014.08.023
- See also: test link — http://dx.doi.org/10.1016/j.joen.2014.02.016